CLINICAL TRIAL: NCT06232902
Title: A Randomized, Double-blind, Single-dose, Parallel-group Study to Compare the Pharmacokinetics and Safety of QL1101 and EU-Avastin® in Healthy Volunteers
Brief Title: A Study to Compare the Pharmacokinetics and Safety of QL1101 and EU-Avastin® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL1101-102
Record Dates: First submitted 2024-01-21; First posted 2024-01-31 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-01

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1101 (Experimental): QL1101, intravenous infusion 90 min (±5min), D1 (Day 1, single dose)
  Interventions: Drug: QL1101
- Avastin® (Active Comparator): Avastin®, intravenous infusion 90 min (±5min), D1 (Day 1, single dose)
  Interventions: Drug: Avastin®

INTERVENTIONS:
Drug: QL1101 — 3mg/kg, single intravenous infusion over 90 min (± 5 min) on first day
  Arms: QL1101
Drug: Avastin® — 3mg/kg, single intravenous infusion over 90 min (± 5 min) on first day
  Arms: Avastin®

SUMMARY:
The goal of this clinical trial is to compare the pharmacokinetic and safety similarity of QL1101 with EU-Avastin® in healthy male volunteers.

Participants will receive a single injection of QL1101/ EU-Avastin®.Researchers will compare pharmacokinetic, safety, and immunogenic similarities between the 2 groups.

DETAILED DESCRIPTION:
This is a phase I,single center, randomized, double-blind and parallel group clinical trial .

The primary objective is to assess the pharmacokinetic similarity of single injections of QL1101 or EU-Avastin® in healthy volunteers.

The secondary objective are to assess the clinical safety and immunogenicity similarity of single injections of QL1101 or EU-Avastin® in healthy volunteers.

Subjects would receive a single 100mg（4ml） of QL1101or EU-Avastin® injection.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily sign the written ICF;
2. Males aged 18- 50 years(inclusive).
3. Body weight between 50.0 kg and 90.0 kg (inclusive), body mass index (BMI) between 18.0 kg/m2 and 28.0 kg/m2 (inclusive);
4. Subjects who agree to practice effective contraception (including but not limited to physical contraception, surgery, or abstinence) throughout the study period until at least 6 months after study drug administration; See Appendix 3 for details;
5. Subjects with no disease history or with a previous medical history which is not clinically significant or has no influence on the study as determined by the study doctor.

Exclusion Criteria:

1. Subjects who have previously suffered or are currently suffering from any clinically significant diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, haematology, immunology and metabolic abnormalities or any other diseases that can interfere with the test results;
2. Abnormalities in clinical laboratory tests, preoperative infectious markers, Chest X-ray, 12-lead ECG, physical examination, vital signs, Abdominal ultrasound were clinically significant or judged to have an impact on the study (based on the judgment of the clinical study doctor);
3. History of hereditary bleeding, thrombophilia, thrombosis (eg, cerebral thrombosis, arteriovenous thrombosis), or history of non-traumatic bleeding and appropriate treatment, or any other condition that may predispose the subject to increased risk of bleeding or thrombosis (eg, thrombocytopenia, or INR > 1.5, etc.);
4. Hypersensitivity to the investigational products or any component of the investigational products, history of specific allergy (Recurrent asthma, urticaria, eczema, etc.) or allergic constitution (such as two or more drugs, food such as milk and pollen allergy);
5. Subjects with a history of gastrointestinal perforation, gastrointestinal fistula or any fistula or inflammatory bowel disease;
6. Recent infection requiring systemic anti-infective treatment within 28 days or serious infection (hospitalization and/or requiring intravenous antibiotics) within 6 months before administration of investigational product;
7. Subjects who have received surgical operation or bone fracture within 4 weeks before screening, or plan to receive surgical operation during the study;
8. One of the HBsAg, hepatitis C antibody, HIV antibody or Treponema pallidum antibody were tested positive;
9. Subjects who have taken any medicine or healthcare product (including Chinese herbal medicine) within 14 days before administration of investigational product;
10. Subjects who have received any biological products or live virus vaccines within 3 months or monoclonal antibodies within 9 months before the study treatment, or bevacizumab or VEGF targeted agents (such as aflibercept, ranibizumab, Conbercept, etc.) before administration of investigational product;
11. Subjects who have participated in the clinical study and administered the investigational product within 3 months before administration of investigational product;
12. Blood donors within 3 months before administration of investigational product;
13. Excessive consumption of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day;
14. Subjects who are addicted to smoking or smoke more than 5 cigarettes per day in the 3 months before screening;
15. Alcoholics or regular drinkers within 6 months before screening, defined as drinking more than 14 units of alcohol per week (1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
16. Drug abusers or those who have used soft drugs (such as marijuana) 3 months before screening or hard drugs (such as cocaine, phencyclidine, etc.) 1 year before screening;
17. Urine drug screening and breath test for alcohol was tested positive before administration of investigational product;
18. Subjects who may not be able to complete this study for other reasons or should not be included in the investigator's opinion.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin® after a single intravenous infusion in healthy volunteers
Cmax | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin® after a single

SECONDARY OUTCOMES:
AUC0-t | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin®
Tmax | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin®
t1/2 | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin®
CL | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin®
Vd | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin®
(AUC0--∞ -AUC0-t)/（AUC0--∞×100%) | 99 day
  To evaluate pharmacokinetic similarity between QL1101 and Avastin®
the rate of treatment-related adverse events as assessed by NCI CTCAE v5.0 | 99 day
  Safety, as defined by the rate of treatment-related adverse events as assessed by NCI CTCAE v5.0.after a single intravenous infusion in healthy volunteers;
immunogenicity | 99 day
  Immunogenicity will be assessed by the incidence of ADA and Nab.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jilin University, Changchun, Jilin, China